CLINICAL TRIAL: NCT07091812
Title: Ultrasonic Vagus Nerve Stimulation: Effectiveness of Blinding and Occurrence of Adverse Effects in Healthy Volunteers
Brief Title: Blinding and Adverse Effects of Ultrasonic Vagus Nerve Stimulation (U-VNS)
Acronym: BLAST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Magdalena Sereda, Assistant Professor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FMHS 29-1124
Record Dates: First submitted 2025-07-11; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: U-VNS; Sham U-VNS
Keywords: tinnitus; vagus nerve stimulation; blinding; adverse effects
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- U-VNS (Experimental): Active ultrasound vagus nerve stimulation
  Interventions: Device: Ultrasound Vagus Nerve Stimulation (U-VNS)
- Sham (Sham Comparator): Sham device indistinguishable from real U-VNS stimulator
  Interventions: Device: Sham U-VNS

INTERVENTIONS:
Device: Ultrasound Vagus Nerve Stimulation (U-VNS) — Ultrasound stimulation of the auricular branch of the vagus nerve using the ZenBud device manufactured by NeurGear (Rochester, New York, USA), a CE-compliant over-the-ear headset. It delivers low-intensity focused ultrasound to the auricular branch of the vagus nerve through several layers of skin (centre frequency 5.3 MHz, pulse repetition rate 41 hertz, 50% duty cycle, average intensity of 1.03 MPa).
  Arms: U-VNS
Device: Sham U-VNS — Sham device, also produced by NeurGear, which is identical in appearance to the true ZenBud device, emits the same sound and warms up slightly where the transducer sits on the skin.
  Arms: Sham

SUMMARY:
The vagus nerve is a large nerve that runs from the gut to the brain. It consists of two main sections, left and right, and comprises a series of branches. One of these branches runs through the ear. Stimulating the vagus nerve with a stimulation device, either implanted in the body or applied to the skin, has been used to treat a number of health conditions associated with the functioning of the vagus nerve. It has also been explored for tinnitus. Tinnitus is the perception of sound in the absence of an external source. It is believed to be related to abnormal activity in the brain. Stimulation of the vagus nerve may be an effective way of normalising this brain activity, thereby reducing tinnitus.

Two types of vagus nerve stimulation (VNS) have been trialled: 1) invasive VNS, using a surgically implanted vagus nerve stimulator and 2) non-invasive VNS, using electrical stimulation devices that are placed on the skin, near a section of the vagus nerve. Past studies of these techniques show that VNS may be a promising future treatment for tinnitus. However, there is not enough data available to draw a firm conclusion on whether VNS is effective at reducing tinnitus or not. Furthermore, all previous studies of VNS for tinnitus have used electrical stimulation of the vagus nerve. Stimulating the vagus nerve, whether through an implanted device or a device on the skin, comes with serious technical challenges. Most importantly, electric currents follow the path of least resistance. When running through biological tissues, such as skin, cartilage or bone, it is difficult to aim for the part of the body that needs to be stimulated. This means it isn't always easy to tell whether the vagus nerve is indeed being stimulated and how much of the current is actually reaching the vagus nerve.

This problem can be overcome by ultrasound stimulation. Ultrasound stimulation employs high frequency sound waves to stimulate tissue. These soundwaves travel through the human body much more predictably than electric currents. As such, ultrasound stimulation of the vagus nerve may be more effective than electrical stimulation. The ZenBud device is designed to apply ultrasound stimulation to part of the vagus nerve that runs through the ear. Ultrasound stimulation allows for more targeted stimulation, increasing the chance of the stimulation reaching the vagus nerve. The ZenBud device is safe for use in healthy adults and received CE marking based on CE assessments conducted at the University of Nottingham Appendix VI-IX).

However, before this device can be used to test whether this approach can reduce tinnitus symptoms, two questions must be answered: Firstly, can people tell whether they're receiving the real VNS or a placebo? Secondly, what are the type, onset and duration of any adverse effects resulting from U-VNS? We know from the testing performed as part of the CE marking that it is safe. However, there may still be mild adverse effects, such as redness, warming up of the skin etc. It is important to understand these mild adverse effects, so that participants can be fully informed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Good general health
* Willing and able to provide informed consent
* Not currently taking any prescribed medication (except contraceptive pill)
* Able and willing to remove any piercings in the ears

Exclusion Criteria:

* Current or past diagnosis of a neurological psychiatric condition
* Current or past diagnosis of cardiac arrhythmia
* Use of medication or recreational drugs that affect the nervous system in the past 3 months
* Currently pregnant
* Allergy to aquasonic gel or any of its components (propylene glycol, glycerin, isothiazolinones)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Effectiveness of blinding and adverse effects questionnaire | Day 1, post-intervention and Day 8, post-intervention
  Questionnaire to assess effectiveness of blinding and characterise adverse effects. Question relating to blinding: participants were asked "Do you believe you received real or sham stimulation?" and given the options Real, Sham, and I don't know to choose from. The responses were used to calculate James' Blinding Index. Adverse effects: participants were asked at the end of each session: "Please indicate the extent to which, if any, you felt the following sensations by using the scale below" followed by a list of possible effects: Itching, Burning, Pain, Tingling, Headache, Warmth/heat, Metallic taste, Fatigue, Nausea, Redness, Other and the rating options None, Mild, Moderate and Severe. Participants were also asked "How long did the sensations last?" with the options It stopped quickly, It stopped around the middle of the session, It stopped around the end of the session and It continued after the end of the session.

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Nottingham BRC Hearing Theme, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data for which consent to share has been obtained will be shared via the University of Nottingham data archive under a CC-BY license. Any data which is deemed to be personally or commercially sensitive will assessed on a case-by-case basis to determine whether it can be shared. There will be no need to update the data past the project period. All published outputs will contain a Data Availability Statement including the datacite DOI that directs to the relevant data set. Data will be released at the same time as any published outputs underpinned by the data or by one year from the end of the project.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be released at the same time as any published outputs underpinned by the data or by one year from the end of the project.